CLINICAL TRIAL: NCT06846476
Title: The Effect of Using Insoles Specially Designed for Diabetic Foot on Postural Balance and Gait Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Yağmur UYSAL, Lecturer, Medipol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedipolU-OPZ-YU-01
Record Dates: First submitted 2025-02-14; First posted 2025-02-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Foot Ulcer (DFU); Orthoses; Postural Balance; Plantar Pressure Distrubution
Keywords: Diabetic Foot; Insole; Postural Balance; Plantar Pressure
MeSH Terms: conditions — Diabetic Foot | interventions — Foot Orthoses; Postural Balance; Oxygen Saturation

STUDY DESIGN:
Intervention Model Description: There will be only one group in our study. This group will be evaluated before and in the 3rd month of insoles use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): Using diabetic insole and will participate in all assessment methods.
  Interventions: Other: Insole; Other: Demographic Information and Anamnesis Form; Other: Pedobarographic analysis; Other: Postural balance; Other: The Foot Functional Index (FFI); Other: Sensory Evaluation; Other: Orthotic Satisfaction Questionnaire- Q-YTKMD (QUEST 2.0); Other: 6 Minute Walk Test (6MWT); Other: Pulse Oximeter Heart Rate and Oxygen Saturation

INTERVENTIONS:
Other: Insole — The production process of the insoles will be produced by Computer Aided Design and Computer Aided Manufacturing (CAD-CAM) method by making plantar pressure analysis and physical evaluation of the individual.
  The insoles will be designed to reduce the load in areas where the pressure is high with off loading technique. The design of the insoles to be produced individually will be made by the researcher (expert orthotist). The materials to be used in the production of insoles will be determined according to the needs of the participant and materials suitable for diabetic individuals will be preferred. In this context; mostly Ethyl Vinyl Acetate (EVA) and materials with cellular air permeability on the upper surface will be used.
Other: Demographic Information and Anamnesis Form — Demographic information and anamnesis form; demographic information of the participant, disease history, physical condition of the foot, skin condition, medications used, allergic status, surgical history, presence of edema, discolouration and temperature increase.
Other: Pedobarographic analysis — Pedobarographic analysis and evaluation of postural balance are widely used by clinicians and researchers to examine the foot structure and to determine the loading patterns of the foot. The data are obtained with electronic sensors placed on the platform where the gait takes place. The sensors are directly connected to the platforms and the computer system programmed to perform foot analysis. With the pedobarography device, pressure distribution data in the foot are obtained in both static and dynamic conditions.
  Foot plantar pressure analysis and postural balance will be performed using the EsCoSCAN® static and dynamic pedobarographic assessment device.
  During the analysis, the individual will be made to stand without moving while looking straight ahead in the standing position for static analysis. This evaluation will be performed before and 3 months after the use of insoles.
Other: Postural balance — Postural balance assessment in the study will be performed with 'Becure Balance System (Becure Global GmbH)'. Individuals will be evaluated for balance on the device with eyes open-closed, single foot-double foot. This evaluation will be performed before and 3 months after the use of insoles.
Other: The Foot Functional Index (FFI) — The Foot Functional Index (FFI) consists of pain, disability and activity limitation and contains a total of 23 items. Pain and disability titles consist of 9 questions each. The pain item measures the severity of foot pain in different situations. The 9 items in the inability heading assess the severity of the difficulty in performing functional activities due to the person's foot problems.
  The activity limitation heading consists of 5 items and measures the activity limitations of the person due to foot problems. AFI is a self-completed scale. Individuals answer the questions with a Visual Analogue Scale (VAS), taking into account their foot condition one week ago. A high score indicates more pain, inability and activity limitation. This evaluation will be performed before and 3 months after the use of insoles.
Other: Sensory Evaluation — Diabetic foot ulcer (DFU), which is one of the microvascular complications of diabetes, frequently occurs in association with loss of protective sensation due to peripheral neuropathy, ischaemia due to peripheral arterial insufficiency, poor foot care and infection. Loss of pressure sensation caused by peripheral nerve damage will be evaluated with 'Semmes Weinstein' monoflaments. The 5.07 nylon monoflament used in the test was produced to bend when 10 g force was applied. This pressure is applied to specific points on the plantar and dorsal aspect of the foot.
  This evaluation will be performed before and 3 months after the use of insoles.
Other: Orthotic Satisfaction Questionnaire- Q-YTKMD (QUEST 2.0) — It is a standardised and widely used questionnaire developed to examine the satisfaction of individuals using orthotics with the device they use. In 2020, a Turkish validity and reliability study was conducted. QUEST 2.0 consists of 12 items. Of these, 8 items question the assistive device and 4 items question service satisfaction. Scale scoring is calculated with a 5-point Likert scale (1=Not satisfied at all, 5=Very satisfied). This evaluation will be performed after the use of insoles.
Other: 6 Minute Walk Test (6MWT) — Participants will walk for 6 minutes at a speed of their choice in a flat and suitable area of 30 metres. The distance walked in 6 minutes will be recorded in metres.
Other: Pulse Oximeter Heart Rate and Oxygen Saturation — Heart rate and oxygen saturation (SpO2) will be recorded by pulse oximetry before and after the 6MWT. The pulse oximeter is a non-invasive device that attaches to a person's fingertip.

SUMMARY:
Postural control and plantar pressure are affected by many parameters in diabetic individuals. It is considered important to examine the relationship between changes in plantar pressure distribution and postural balance, physiological expenditure index and gait parameters in diabetic individuals. Within the scope of this project, based on the above mentioned reasons, we plan to produce a personalised off loading insoles designed for diabetic foot.

DETAILED DESCRIPTION:
Excessive localized loading on the plantar surface leads to repeated microtrauma and the development of diabetic foot ulcers. The plantar region, subjected to constant weight-bearing pressure, develops chronic wounds due to dangerous vascularity. Excessive plantar pressure is considered the primary risk factor for plantar ulcers in diabetic individuals; custom insoles are considered the gold standard in treatment for off-loading plantar pressure.

The off-loading technique, which reduces plantar pressure, is an effective ulcer prevention strategy for neuropathic feet with impaired sensation and increased plantar load and tissue stress.

A review of the literature shows that previous studies have clearly demonstrated that off-loading insoles are effective in reducing abnormal plantar pressure in a specific area and that they also have some effect on the pressure distribution in surrounding areas. However, the potential impact of this positive effect on postural balance, postural control, and individuals' physiological expenditure and energy consumption has not been sufficiently studied.

Therefore, it is considered important to investigate the relationship between changes in plantar pressure distribution, postural balance, physiological expenditure index, and walking parameters in diabetic individuals.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 40 and 65,
* Wagner Classification stages 0 or 1,
* He has type I or type II diabetes,
* No history of amputation surgery,
* Individuals using shoes suitable for insoles will be included in the study.

Exclusion Criteria:

* - Using an assistive device (long-walking device, walker, canadiene, etc.),
* He has a history of amputation,
* He has a Charcot foot deformity,
* The one with the open wound,
* Physical disability that may restrict joint movement,
* Individuals using shoes that are not suitable for insoles will not be included in the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Postural Balance | the evaluation of balance and postural control will be carried out before and in the 3rd month of insoles use and the effects on individuals will be compared.
  Postural balance assessment in the study will be performed with 'Becure Balance System (Becure Global GmbH)'. It is planned to perform balance assessment of individuals on the device with eyes open-closed, single foot-double foot. After the participant is positioned on the balance board, balance evaluations will be made in different situations such as eyes open-closed, single foot-double foot. Changes in the centre of gravity on the x and y axes with the eyes open and closed, and changes in postural oscillation will be examined with the results of the distance of movement expressing the changes in the centre of gravity. The postural balance assessment conducted in the study provides all the parameters mentioned above in centimeters. These values represent postural sway.

SECONDARY OUTCOMES:
The Physiological Cost Index (PCI) | Evaluation will be made before and in the 3rd month of insoles use.
  A simple and practical method for assessing walking efficiency and energy expenditure. These 3 measurements are obtained during the walking test; PCI = (Working HR - Resting HR) / Walking speed. The physiological expenditure index value reflects increased heart rate. In our project; PCI will be assessed with the 6 Minute Walk Test (6MWT).
  (Heart rate and oxygen saturation (SpO2) will be recorded by pulse oximetry)

CONTACTS AND LOCATIONS:
Overall Officials: YAGMUR UYSAL, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Not sure